CLINICAL TRIAL: NCT00003498
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Patients With Non-Hodgkin's Lymphoma
Brief Title: Antineoplaston Therapy in Treating Patients With Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066537; BC-LY-3 (Other: Burzynski Research Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2020-12-19 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Non Hodgkin Lymphoma
Keywords: Non Hodgkin Lymphoma Recurrent; Non Hodgkin Lymphoma Refractory
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Patients with Non-Hodgkin's Lymphoma will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
Current therapies for Non-Hodgkin's Lymphoma provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of Non-Hodgkin's Lymphoma.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on patients with Non-Hodgkin's Lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and possible effectiveness of antineoplastons A10 and AS2-1 in patients with non-Hodgkin's lymphoma who have failed high-dose chemotherapy and bone marrow transplantation.
* Describe the response to, tolerance to, and side effects of this regimen in these patients.

Non-Hodgkin's Lymphoma patients receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues up to 12 months in the absence of disease progression or unacceptable toxicity.

OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in patients with Non-Hodgkin's Lymphoma, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in patients with Non-Hodgkin's Lymphoma.
* To determine objective response, tumor size is measured utilizing physical examination, radiologic studies, and bone marrow biopsies as necessary, performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven non-Hodgkin's disease that has failed both prior high-dose chemotherapy and bone marrow transplantation

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC greater than 2,000/mm^3
* Platelet count greater than 20,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulatory agents (e.g., interferon or interleukin-2)

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered

Endocrine therapy:

* At least 4 weeks since prior corticosteroids
* No concurrent corticosteroids

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No prior antineoplaston therapy
* No other concurrent antineoplastic agents
* No concurrent antibiotics, antifungals, or antivirals

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 1997-10-13 (Actual); Primary Completion 2007-02-02 (Actual); Study Completion 2007-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Antineoplaston therapy (Atengenal + Astugenal): Patients with Non-Hodgkin's Lymphoma will receive Antineoplaston therapy (Atengenal + Astugenal).
  The daily doses of A10 and AS2-1 are divided into six infusions, which are given at 4-hourly intervals. Each infusion starts with infusion of A10 and is immediately followed by infusion of AS2-1.
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 5
Completed | 1
Not Completed | 4
Not completed — Not evaluable. | 4

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 46.3 [32.3 to 63.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Objective Response, Stable Disease, or Progressive Disease
Description: An objective response is defined as a complete or partial response. A complete response is complete disappearance of all tumor by physical examination and radiographic studies and bone marrow involvement, if appropriate, for a minimum of four weeks. A partial response is a > 50% reduction in the sum of the products of the greatest perpendicular diameters of all measurable lesions compared to the corresponding baseline evaluation, for a minimum of four weeks. Stable disease indicates < 50% change in the sum of the products of the greatest perpendicular diameters of all measurable lesions compared to the corresponding baseline evaluation, for a minimum of twelve weeks. Progressive Disease is a > 50% increase in the sum of the products of the greatest perpendicular diameters of all measurable lesions compared to the corresponding baseline evaluation, for a minimum of four weeks.
Time Frame: 5 months
Measure: Number; unit: participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 1
participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 0
  Progressive Disease | 1

ADVERSE EVENTS:
Time Frame: 9 years, 4 months
Description: Five patients were recruited between October 1997 and January 2007. All study subjects were seen at the Burzynski Clinic in Houston TX
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=5)
Hemorrhage/Bleeding - Other (Inguinal region) (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=5)
Hemoglobin (Blood and lymphatic system disorders) | 3
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Edema/Fluid retention (Skin and subcutaneous tissue disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hemorrhage, GU: Bladder (Renal and urinary disorders) | 1
Hemorrhage/Bleeding - Other (Inguinal region) (Skin and subcutaneous tissue disorders) | 1
Albumin, serum-low (hypoalbuminemia) (Investigations) | 1
Alkaline phosphatase (Investigations) | 2
Hyperbilirubinemia (Investigations) | 1
Hyperglycemia (Investigations) | 1
Hypernatremia (Investigations) | 2
Hypocalcemia (Investigations) | 1
Hypokalemia (Investigations) | 5
Hypomagnesemia (Investigations) | 1
Proteinuria (Investigations) | 1
SGOT (Investigations) | 1
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 1
Tremor (Nervous system disorders) | 1
Pain: Head/headache (General disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No